CLINICAL TRIAL: NCT03335813
Title: Endoesophageal Brachytherapy for Patients With Esophageal Cancer: A Balloon Repositioning, Multichannel Radiation Applicator for Optimizing Treatment Delivery
Brief Title: Endoesophageal Brachytherapy for Patients With Esophageal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE5217
Record Dates: First submitted 2017-11-03; First posted 2017-11-08 (Actual); Results first posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-05

CONDITIONS: Esophageal Cancer
Keywords: brachytherapy; multichannel balloon applicator
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- brachytherapy with multichannel balloon applicator (Experimental): 6 channel balloon re-positioning, multichannel brachytherapy applicator used to deliver localized radiation therapy to esophageal tumors
  Interventions: Device: Endoesophageal Brachytherapy

INTERVENTIONS:
Device: Endoesophageal Brachytherapy — Balloon repositioning, multichannel brachytherapy applicator which has 6 channels instead of 3-tubes which will be used to deliver localized radiation

SUMMARY:
Depending upon the cancer stage, esophageal cancer can be treated with surgery, chemotherapy, radiation therapy, or a combination of these modalities. Sometimes in addition to external radiation therapy or instead of external radiation therapy, select patients with esophageal cancer may benefit from localized radiation to the tumor, called esophageal brachytherapy. There are many different radiation techniques and delivery approaches for this type of specialized radiation therapy, and the purpose of this document is to provide a written summary of an innovative delivery method.

DETAILED DESCRIPTION:
Primary Objective Pilot study of multichannel endoesophageal brachytherapy applicator to determine dose distribution and conformality of a 6 channel balloon repositioning applicator.

Secondary Objective(s)

1. To collect data in order to show how the 6-tube endoesophageal brachytherapy technique will be an improvement (more conformed dose distribution) over a previously designed 3-tube endoesophageal brachytherapy technique in patients who are candidates for esophageal brachytherapy
2. To evaluate acute toxicity of novel endoesophageal brachytherapy applicator.

Study Design

This innovative study will be an improvement over a previously designed 3-tube endoesophageal brachytherapy technique in patients who are candidates for esophageal brachytherapy. The brachytherapy planning process will utilize a novel multichannel balloon applicator.

The initial treatment session will occur after the patient has been found to be eligible, the consent form has been completed, and the treatment plan has been created. The patient will undergo subsequent weekly treatments for 3 to 6 weeks after the initial treatment.

The subject will be expected to participate in the trial throughout its entirety. The participation period is 6 months of which the patient will be evaluated and seen at months 3 and 6.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proved esophageal adenocarcinoma or squamous cell carcinoma
* Disease that can be encompassed in the radiotherapy treatment field
* Women of childbearing potential must practice adequate contraception
* Subjects must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Concurrent chemotherapy at the time of brachytherapy treatments
* Tracheal or bronchial involvement
* Cervical esophagus location
* Stenosis that cannot be bypassed or dilated to allow for applicator placement
* Not willing or unable to provide informed consent
* History of esophageal fistula

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2020-11-14 (Actual); Study Completion 2020-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John F Greskovich, MD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Weston, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Brachytherapy With Multichannel Balloon Applicator
Started | 7
Completed | 6
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Brachytherapy With Multichannel Balloon Applicator
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Dose of Radiation Delivered to 90% of Tumor Volume (D90)
Description: Percent of prescription dose received by 90% of PTV (planning target volume)
Time Frame: Up to 6 months of follow-up
Population: Number of participants who received treatment
Measure: Median (Full Range); unit: percentage of Prescription dose
Arm/Group | Brachytherapy With Multichannel Balloon Applicator
Number analyzed (Participants) | 6
percentage of Prescription dose | 105.5 [69.84 to 115.34]

2. Primary Outcome: Percent Volume of the Tumor Receiving the Prescription Dose (V100)
Description: Percent volume of the tumor receiving 100% of the prescription dose calculated as the mean from the total weekly HDR brachytherapy treatment plans
Time Frame: Up to 6 months of follow-up
Population: Number of participants who received treatment
Measure: Mean (Full Range); unit: percentage of volume
Arm/Group | Brachytherapy With Multichannel Balloon Applicator
Number analyzed (Participants) | 6
percentage of volume | 94.3 [66.0 to 97.9]

3. Secondary Outcome: Radiation Treatment Volume
Description: Volume of tissue, both tumor plus normal tissue volume, receiving 100% of the prescription dose
Time Frame: Up to 6 cycles (6 weeks) of treatment
Population: Number of Participants who received treatment
Measure: Median (Full Range); unit: cc
Arm/Group | Brachytherapy With Multichannel Balloon Applicator
Number analyzed (Participants) | 6
cc | 52.13 [38.93 to 90.40]

4. Secondary Outcome: Dose of Radiation to Organ at Risk (Bronchus)
Description: Dose to 1cc volume of the trachea-mainstem bronchus calculated as the mean dose from the total weekly HDR brachytherapy treatment plans for the 4 participants who had tumors in proximity to the trachea or mainstem bronchus.
Time Frame: Up to 6 months of follow-up
Population: Number of Participants who had tumors in proximity to the specified organ
Measure: Median (Full Range); unit: Gy
Arm/Group | Brachytherapy With Multichannel Balloon Applicator
Number analyzed (Participants) | 4
Gy | 2.38 [.76 to 3.79]

5. Secondary Outcome: Dose of Radiation to Organ at Risk (Heart)
Description: Dose to 1 cc volume of the heart calculated as the mean dose from the total weekly HDR brachytherapy treatment plans for the 4 participants who had tumors in proximity to the heart.
Time Frame: Up to 6 months of follow-up
Population: Number of Participants who had tumors in proximity to the specified organ
Measure: Median (Full Range); unit: Gy
Arm/Group | Brachytherapy With Multichannel Balloon Applicator
Number analyzed (Participants) | 4
Gy | 3.22 [2.44 to 4.18]

6. Secondary Outcome: Dose of Radiation to Organ at Risk (Aorta)
Description: Dose to 1 cc volume of the aorta calculated as the mean dose from the total weekly HDR brachytherapy treatment plans for the 6 participants who had tumors in proximity to the aorta.
Time Frame: Up to 6 months of follow-up
Population: Number of Participants who had tumors in proximity to the specified organ
Measure: Median (Full Range); unit: Gy
Arm/Group | Brachytherapy With Multichannel Balloon Applicator
Number analyzed (Participants) | 6
Gy | 3.19 [1.86 to 5.62]

7. Secondary Outcome: Tumor Response Based on Resist Criteria
Description: Tumor response determined by endoscopic evaluation of tumor at time of last brachytherapy treatment. Endoscopic CR is defined as no visible tumor at end of treatment -on endoscopy exam and PR is defined as a persistent tumor at the end of treatment.
Time Frame: Up to 6 months of follow-up
Population: All Participants who received treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Brachytherapy With Multichannel Balloon Applicator
Number analyzed (Participants) | 6
Participants
  Endoscopic CR | 5
  Endoscopic PR | 1

8. Secondary Outcome: Number of Participants With Esophageal Ulceration
Description: Presence of an ulceration of the mucosa in area of brachytherapy treatment
Time Frame: Up to 6 cycles (6 weeks) of treatment
Population: All Participants who received treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Brachytherapy With Multichannel Balloon Applicator
Number analyzed (Participants) | 6
Participants | 5

9. Secondary Outcome: Number of Participants With Esophageal Fistula
Description: Presence of a fistula between the esophagus and trachea, mainstem bronchus or mediastinum
Time Frame: Up to 6 cycles (6 weeks) of treatment
Population: All Participants who received treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Brachytherapy With Multichannel Balloon Applicator
Number analyzed (Participants) | 6
Participants | 0

10. Secondary Outcome: Number of Particiapants With Esophageal Stricture
Description: Presence of an esophageal stricture
Time Frame: Up to 6 cycles (6 weeks) of treatment
Population: All Participants who received treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Brachytherapy With Multichannel Balloon Applicator
Number analyzed (Participants) | 6
Participants | 3

11. Secondary Outcome: Number of Participants With the Need for Dilation
Description: Number of participants with the need for esophageal dilation
Time Frame: Up to 6 cycles (6 weeks) of treatment
Population: All participants who received treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Brachytherapy With Multichannel Balloon Applicator
Number analyzed (Participants) | 6
Participants | 3

12. Post Hoc Outcome: Number of Participants With Need for Stent Placement
Description: Need for esophageal stent
Time Frame: Up to 6 cycles (6 weeks) of treatment
Population: Number of participants who received treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Brachytherapy With Multichannel Balloon Applicator
Number analyzed (Participants) | 6
Participants | 2

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Brachytherapy With Multichannel Balloon Applicator
All-Cause Mortality (participants affected / at risk) | 5/7
Serious Adverse Events (participants affected / at risk) | 5/7
Other Adverse Events (participants affected / at risk) | 0/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brachytherapy With Multichannel Balloon Applicator (N=7)
Death, NOS (General disorders) | 1 — disease progression and pneumonia
Death, NOS (General disorders) | 1 — disease progression with neutropenic fevers, RLL pneumonia, and sepsis
Death, NOS (General disorders) | 1 — hospice progressive weakness
Death, NOS (General disorders) | 1 — overall poor prognosis
Death, NOS (General disorders) | 1 — Due to intestinal issues

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-22): https://cdn.clinicaltrials.gov/large-docs/13/NCT03335813/Prot_SAP_002.pdf
  • Informed Consent Form (2017-11-22): https://cdn.clinicaltrials.gov/large-docs/13/NCT03335813/ICF_003.pdf